CLINICAL TRIAL: NCT05114564
Title: Evaluation of the Performance of Monthly Replacement Sphere Lens Designs in Habitual Soft Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-129
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Results first posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A, Then Lens B (Experimental): Participants will wear Lens A for one month and then cross over to wear Lens B for one month.
  Interventions: Device: Lens A (comfilcon A lens); Device: Lens B (lehfilcon A lens)
- Lens B, Then Lens A (Experimental): Participants will wear Lens B for one month and then cross over to wear Lens A for one month.
  Interventions: Device: Lens A (comfilcon A lens); Device: Lens B (lehfilcon A lens)

INTERVENTIONS:
Device: Lens A (comfilcon A lens) — 1 month
Device: Lens B (lehfilcon A lens) — 1 month

SUMMARY:
The objective of the study is to evaluate the clinical performance of two monthly silicone hydrogel contact lenses in habitual wearers of frequent replacement (FRP) lenses when worn for one month.

DETAILED DESCRIPTION:
This study is a prospective, bilateral eye, double-masked, randomized, 1-month cross-over, daily-wear design involving two different FRP lens types. Each lens type will be worn for approximately one month.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age and no older than 35 years, and has full legal capacity to volunteer;
* Has read and signed an information consent letter;
* Is willing and able to follow instructions and maintain the appointment schedule;
* Self-reports having a full eye examination in the previous two years;
* Self-reports spending on most days at least 6 hours cumulative (not necessarily in one single stretch) using digital devices such as a computer, laptop, tablet, e-reader, smartphone;
* Has healthy eyes with no health condition or medication that contra-indicate contact lens wear, in the opinion of the investigator;
* Anticipates being able to wear the study lenses for at least 8 hours a day, 6 days a week;
* Habitually wears soft frequent replacement contact lenses, for the past 3 months minimum (NOTE: the habitual contact lens brand is restricted such that no more than one third are to be the Biofinity brand (or their equivalent private label brand name) and no more than one third are to be an Alcon brand;
* Has refractive astigmatism no higher than -0.75DC in each eye;
* Can be fit and achieve binocular distance vision of at least 20/30 Snellen (Available lens parameters are sphere +6.00 to -6.00D, 0.25D steps).

Exclusion Criteria:

* Is participating in any concurrent clinical or research study;
* Has any known active ocular disease and/or infection that contraindicates contact lens wear;
* Has a systemic or ocular condition that in the opinion of the investigator may affect a study outcome variable;
* Is using any systemic or topical medications that in the opinion of the investigator may affect contact lens wear or a study outcome variable;
* Has known sensitivity to the diagnostic sodium fluorescein used in the study;
* Self-reports as pregnant, lactating or planning a pregnancy at the time of enrolment;
* Has undergone refractive error surgery or intraocular surgery.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD FCOptom, Study Director — Centre for Ocular Research and Education
Locations (4):
- United States (4):
  - Complete Eye Care of Medina, Medina, Minnesota
  - Sacco Eye Group, Vestal, New York
  - Athens Eye Care, Athens, Ohio
  - ProCare Vision Center, Granville, Ohio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty-six participants were screened. Of the 66 that were dispensed with lenses, two were discontinued.
  One of the completing participants presented at the final visit wearing an unknown lens. It was decided to exclude all the data for this participant and this finding was reported as a major protocol deviation. All remaining participants who completed the study were included in the analysis (Analysis population n=63).
Groups:
- Lens B, Then Lens A: Participants wore Lens B for one month and then crossed over to wear Lens A for one month.
- Lens A, Then Lens B: Participants wore Lens A for one month and then crossed over to wear Lens B for one month.
Period: First Intervention
Arm/Group | Lens B, Then Lens A | Lens A, Then Lens B
Started | 34 | 32
Completed | 33 | 31
Not Completed | 1 | 1
Not completed — Vision with study contact lens subjectively unacceptable | 1 | 0
Not completed — Adverse Event | 0 | 1
Period: Second Intervention
Arm/Group | Lens B, Then Lens A | Lens A, Then Lens B
Started | 33 | 31
Completed | 33 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Sixty-six participants were screened, and demographic data include all screened participants.
Groups:
- Overall Study: Total study population
Arm/Group | Overall Study
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subjective Ratings on Lens Handling on Removal
Description: Subjective Ratings on Lens handling on removal (0-10 scale, 0.5 steps; 10=very easy, 0=very difficult)
Time Frame: Day 27
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lens A: Participants wore Lens A for one month.
- Lens B: Participants wore Lens B for one month.
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 63 | 63
units on a scale | 8.6 (1.6) | 8.5 (2.2)

ADVERSE EVENTS:
Time Frame: From dispense up to one month on each study lens, for a total of two months
Arm/Group | Lens A | Lens B
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 3/66 | 2/66
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lens A (N=66) | Lens B (N=66)
COVID-19 (Social circumstances) | 2 | 1
Sinus infection (Infections and infestations) | 0 | 1
Single infiltrate in superior cornea (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT05114564/Prot_SAP_000.pdf